CLINICAL TRIAL: NCT03311971
Title: Single Center Study Evaluating the Possible Effect of Virtual Reality Spectacles on Pain Following Total Knee Replacement Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, DROR ROBINSON, Head of orthopedic research unit, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0428-17-RMC
Record Dates: First submitted 2017-08-30; First posted 2017-10-17 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Pain Post Joint Arthroplasty

STUDY DESIGN:
Intervention Model Description: Comparison of intervention with conventional therapy. The intervention group includes use of virtual reality spectacles. The control group includes routine postoperative care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (Sham Comparator): Patient undergoing conventional analgesic therapy after total knee replacement
  Interventions: Device: No VR glasses
- Virtual reality glasses (Experimental): Patient undergoing conventional analgesic therapy after total knee replacement and treated with virtual glasses
  Interventions: Device: Virtual reality glasses

INTERVENTIONS:
Device: Virtual reality glasses — Patients will be treated with virtual glasses
  Arms: Virtual reality glasses
Device: No VR glasses — Patients will not use VR glasses
  Arms: Conventional therapy

SUMMARY:
The trial aims to evaulate the possiblity that use of virtual reality spectacles will affect post operative pain in total knee arthroplasty patients. The trial is a single center open label design. Patients will be randomized into two arm study comparing the effect of the use of virtual reality spectacles on pain levels and analgesic consumption in the perioperative period. The controls shall receive standard post operative care. The endpoints are VAS levels and analgesic use.

DETAILED DESCRIPTION:
Evaluation Procedure This is a single center, interventional, randomized, unblinded two arm study assessing pain and analgesic use in post knee arthroplasty patients. The randomization ratio is 2:1 intervention to control. Both groups will receive routine post operative care. The intervention group will be treated with virtual reality spectacles. The control group will receive routine post operative care. Pain levels will be assessed using VAS and analgesic use.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee arthroplasty gender indifferent, aged over 18 years old
* Patient with ability to see in three dimensions

Exclusion Criteria:

* Inability to comply with the study protocol
* Single eye vision
* Blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
VAS pain response | One week
  questionnaires

SECONDARY OUTCOMES:
Analgesic use | one week
  amount of analgesic medication consumed

CONTACTS AND LOCATIONS:
Locations (1):
- Hasharon Hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No